CLINICAL TRIAL: NCT02605252
Title: A Study on Optimizing HBsAg Clearance in CHB Patients With Sequential Treatment of Pegylated Interferon Alpha-2b and Nucleoside Analogues
Brief Title: New Strategy Study of Functional Cure of Chronic Hepatitis B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiang Zhu, Attending Physician, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3rd-sysu-hbv-functional cure
Record Dates: First submitted 2015-11-08; First posted 2015-11-16 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic hepatitis B; Peginterferon alfa-2b; Nucleotide analogue
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CHB patients (Experimental): Hepatitis B e antigen (HBeAg)-negative CHB patients who had received NAs for more than 12 months, with HBsAg <1500 IU/ mL and Hepatitis B virus DNA not detectable, are to receive peginterferon alfa-2b 80 micrograms/week for 48 weeks.
  Interventions: Drug: Peginterferon alfa-2b

INTERVENTIONS:
Drug: Peginterferon alfa-2b — peginterferon alfa-2b 80 micrograms/week for 48 weeks

SUMMARY:
As HBsAg clearance is uncommon in chronic hepatitis B (CHB) patients on nucleoside analogues (NAs) therapy. The purpose of this study is to optimize HBsAg clearance in CHB Patients with sequential treatment of pegylated interferon alpha-2b and NAs.

DETAILED DESCRIPTION:
CHB Patients who had received, and responded to, NAs for more than 12 months are switched to receive peginterferon alfa-2b 80 micrograms/week for 48 weeks and follow up for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. CHB patients who had received NAs for more than 12 months.
2. Hepatitis B e antigen (HBeAg)-negative and anti-HBeAg positive.
3. Hepatitis B surface antigen (HBsAg) positive and <1500 IU/mL.
4. Hepatitis B virus DNA not detectable.

Exclusion Criteria:

1. Patients with liver cirrhosis, Hepatocellular Carcinoma or other malignancies.
2. Patients with other factors causing liver diseases.
3. Pregnant and lactating women.
4. Patients with concomitant HIV infection or congenital immune deficiency diseases.
5. Patients with diabetes, autoimmune diseases.
6. Patients with important organ dysfunctions.
7. Patients with serious complications ( e.g., infection, hepatic encephalopathy, hepatorenal syndrome, gastrointestinal bleeding. )
8. Patients who receive antineoplastic or immunomodulatory therapy in the past 12 months.
9. Patients who can't come back to clinic for follow-up on schedule.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
HBsAg loss | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Zhu, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The third affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No